CLINICAL TRIAL: NCT06090032
Title: Copmined Sono-pulmonary Score and APACHE Score as a Predictor of Outcome in Respiratory Intensive Care Unit Patients With Ventilator Associated Pneumonia
Brief Title: Compined SONOPULMONARY Infection Score and APACHE Score in RICU Patients With VAP
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Lamiaa Hussein Fouda, Doctor, Assiut University
Other Study IDs: Chest U/S in RICU PT WITH VAP
Record Dates: First submitted 2023-10-13; First posted 2023-10-19 (Actual); Last update posted 2023-10-19 (Actual); Status verified 2023-10

CONDITIONS: Respiratory Intensive Care Unit Patients With Ventilator Associated Pneumonia
MeSH Terms: interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Ultrasound — We will use ultrasongraphy as a part of assessment in respiratory intensive care unit patients with ventilator associated pneumonia

SUMMARY:
Aim of the study :

1. Efficacy of Sono pulmonary infection score in combination with APACHE score in early diagnosis of VAP
2. Assessment of prediction role of combined SIPS SCORE and APACHE SCORE of outcome of VAP patient in RICU
3. Assessments of role of ultrasonography in early diagnosis and follow up of VAP

DETAILED DESCRIPTION:
Pneumonia is a bacterial, viral or fungal infection of the lungs, which causes the alveoli of the lungs to fill up with microorganisms, fluid and inflammatory cells, preventing the lungs from functioning effectively[1]. Ventilator associated pneumonia (VAP) is the most common and a leading cause of death in intensive care unit patient. Ventilator associated pneumonia is caused by prolonged duration of mechanical ventilation ,and prolonged hospital stay, which increase hospital costs, possibly increase mortality rate, and increase antibiotic use in ICU patients , early identification of VAP is an important clinical goal to improve patient outcomes [2]. In recent year several scoring systems have been developed to evaluate the severity of illness and to predict the outcome, especially the mortality rate of intensive care unit patient, such as the Clinical pulmonary infection score (CPIS) or modified (CPIS)The Clinical Pulmonary Infection Score (CPIS) was developed to serves a tool to facilitate the diagnosis of ventilator-associated pneumonia (VAP),The CPIS is calculated on the basis of points assigned for various signs and symptoms of pneumonia (eg, fever and extent of oxygenation mpairment) ,a CPIS has an average between 0-12>6 some studies suggest that CPIS >6 may correlate with VAP Sonar is easy bedside test to diagnose pleural effusion, pneumonia pneumothorax , so recently lung ultrasonography (LUS) incorporated in evaluation and diagnosis of VAP in a new score called sono pulmonary infection score (SPIS) . The (SPIS), where is incorporated LUS finding instead of CXR finding of CPIS is assigned two points for ≥ one area of dynamic air bronchogram. One point was given for ≥ two sub-pleural consolidation or lobar consolidation areas or ≥ one sub-pleural, and ≥one lobar consolidationRecently (combination of SPIS with APACHE score in assessment of VAP is under research ).

ELIGIBILITY:
Inclusion Criteria:

1. Age >18 yrs
2. Mechanically ventilated patients after first 48 hours of admission in RICU

Exclusion Criteria:

1. Age <18 yrs
2. Patients already diagnosed pneumonia
3. Malignancy
4. patient refused participation in the study.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Mechanically ventilated patients after first 48 hours of admission in RICU .
Sampling Method: Non-Probability Sample
Enrollment: 53 (Estimated)
Dates: Start 2023-11-01 (Estimated); Primary Completion 2024-11-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Compined SONOPULMONARY infection score and APACHE score as a predictor of outcome in RICU patients with ventilator associated pneumonia | One year
  Compined SONOPULMONARY infection score and APACHE score as a predictor of outcome of respiratory intensive care unit patients with ventilator associated pneumonia

REFERENCES:
- See also: The National Institute for Health and Care Excellence (NICE), Pneumonia in adults: diagnosis and management. 2019 — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC8830125/
- See also: 3. (Klevens RM, Edwards JR, Richards CL, et al. Estimating health careassociated infections and deaths in U.S. hospitals, 2002, Public Health Rep, 2007, vol. 122 (pg. 160-166). — https://pubmed.ncbi.nlm.nih.gov/20597663/
- See also: 4. Mongodi S, Via G, Girard M, Rouquette I, Misset B, Braschi A et al. Lung ultrasound for early diagnosis of ventilator-associated pneumonia. Chest. 2016;;149((4):969--980.. doi: 10.1016/j.chest.2015.12.012 — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC7991773/
- See also: . Knaus WA, Zimmerman JE, Wagner DP, Draper EA, Lawrence DE. APACHE-acute physiology and chronic health evaluation: A physiologically based classification system. Crit Care Med. 1981;9:591-7. — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC8225448/